CLINICAL TRIAL: NCT04928274
Title: Evaluation of Bone Height Changes In Three Implants Retained Mandibular Overdenture Using Three Different Attachment Design. A Randomized Clinical Trial.
Brief Title: Bone Height Changes In Three Implants Retained Mandibular Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Ragheb, Lecturer , Prosthodontist, Department of Prosthodontics, Faculty of Oral & Dental Medicine,Kafr El-shiekh University, Kafr El-shiekh ,Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KD/11/21
Record Dates: First submitted 2021-06-04; First posted 2021-06-16 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Bone Loss; Implant Site Reaction
Keywords: implant - over denture - bone height changes - attachment
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded operators have carried out the assessment of bone height changes in order to have accurate results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ball retained mandibular over denture (Other): each patient in this group received 3 implant installed in mandible and 3 ball attachments for retention of over denture
  Interventions: Other: ball attachment to retain mandibular over denture
- locator retained mandibular over denture (Other)
  Interventions: Other: locator attachment to retain mandibular over denture
- telescopic retained mandibular over denture (Other)
  Interventions: Other: telescopic attachment to retain mandibular over denture

INTERVENTIONS:
Other: ball attachment to retain mandibular over denture — each patient in group receive 3 locator attachment for over denture retention
  Arms: ball retained mandibular over denture
Other: locator attachment to retain mandibular over denture — each patient in group receive 3 locator attachment for over denture retention
  Arms: locator retained mandibular over denture
Other: telescopic attachment to retain mandibular over denture — each patient in group receive 3 telescopic attachment for over denture retention
  Arms: telescopic retained mandibular over denture

SUMMARY:
this study was to compare the bone height changes around three implant telescopic, locator, and ball retained mandibular overdentures. radiographic changes in peri-implant tissue in three groups were evaluated

DETAILED DESCRIPTION:
Twenty-four completely edentulous patients were recruited from the outpatient clinic of Removable Prosthodontics Cairo University. All patients recruited were seeking to install implants in their lower jaw, and have to meet the following inclusion criteria: age ranging from 50 to 69 years old, patients should have no contra-indication for implant installation, all patients should perform a glycosylated hemoglobin analysis and only up to 8 were included in the study. All patients had to sign an informed consent before the start of the study, and have to comply with the assigned follow-ups. Patients with any contraindications for implant placement or those who didn't comply with the follow ups were excluded from the study.

All patients included had maxillary and mandibular complete dentures fabricated following the conventional steps, after a period of 6 weeks adaptation, all patients were ready for implant installation. The lower denture was duplicated into a radiographic stent, having radio-opaque markers in the areas of implant installation. All patients had a CBCT x ray wearing the radiographic stent, to allow for proper implant planning and to visualize the height and width of the osteotomy site. The radiographic stent was then modified to a surgical stent by making a tunnel corresponding to the site of implant installation. All Patients in this study received three implants in the lower jaw at the premolar-canine area bilaterally and one implant in the midline at the central incisor area.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 50 to 69 years old, patients should have no contra-indication for implant installation, all patients should perform a glycosylated hemoglobin analysis and only up to 8 were included in the study

Exclusion Criteria:

* Patients with any contraindications for implant placement or those who didn't comply with the follow ups were excluded from the study.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Bone height measurement | one year
  The Digora software was then used to measure bone height changes on the mesial and distal surface of each implant. The Digora software was then used to measure bone height changes on the mesial and distal surface of each implant. The implant in the peri-apical x ray was calibrated by drawing a line from the junction of the implant and abutment to the apical end of the implant, this line was the calibration line corresponding to the implant real length which was 11.5mm. After the implant was calibrated, a line was drawn on each implant surface; at the mesial and distal surface starting from the first implant thread to bone contact to the apical implant thread to bone contact. The line drawn would correspond to the bone height on each surface . Two blinded operators have carried out the assessment of bone height changes in order to have accurate results.

CONTACTS AND LOCATIONS:
Overall Officials: Nouran Abdel Nabi, phd, Principal Investigator — Cairo University
Locations (3):
- Egypt (3):
  - Faculty of Dentistry , Kafrelshiekh university, Kafr ash Shaykh, Kafr el-Sheikh Governorate
  - Cairo University, Cairo
  - Faculty of Dentistry , Kafr El Shiekh University, Kafr ash Shaykh

IPD SHARING:
Plan to Share IPD: No
study protocol